CLINICAL TRIAL: NCT04417179
Title: The Feasibility and Efficacy of Erector Spinae Block Versus Transversus Abdominis Plane Block In Laparoscopic Bariatric Surgery
Brief Title: Erector Spinae Block Versus Transversus Abdominis Plane Block In Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed abdelghany ali, Anesthesia lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD-250-2020
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Erector Spinae Block; Bariatric Surgery Candidate
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block group (Experimental): the TAP block will be given by a high frequency linear ultrasound transducer of Siemens acuson x300 3-5MHz ultrasound .
  a blunted tip , 20-gauge, short bevel needle (Pajunk Sonoplex, Geisingen, Germany) will be used under direct ultrasound visualization, . After confirming the correct placement of the needle and the negative aspiration probe anaesthetic substance will be injected along the subcostal line in the transversus abdominis plane 20 ml 0.25% bupivacaine(10) , and the dissection of the plane was observed. The block will be performed bilaterally.
  Interventions: Procedure: transversus abdominis block; Drug: Bupivacaine 0.25% Injectable Solution; Device: Siemens Acuson x300 3-5MHz Ultrasound
- ESP group (Experimental): the Erector Spinae block will be given by a high-frequency linear ultrasound transducer of Siemens acuson x300 3-5MHz ultrasound .A blunted tip , 20-gauge, short bevel needle (Pajunk Sonoplex, Geisingen, Germany) will be used under strict aseptic precautions until the tip is deep to erector spinae muscle, The block will be performed bilaterally by injecting 40 mL of 0.25% bupivacaine (20 mL into each side) into the fascial plane between the deep surface of the Erector Spinae muscle and the transverse processes of the lumbar vertebrae laterally
  Interventions: Procedure: Erector spinae block; Drug: Bupivacaine 0.25% Injectable Solution; Device: Siemens Acuson x300 3-5MHz Ultrasound

INTERVENTIONS:
Procedure: transversus abdominis block — transversus abdominis block
  Arms: TAP block group
Procedure: Erector spinae block — Erector spinae block
  Arms: ESP group
Drug: Bupivacaine 0.25% Injectable Solution — Local Anesthetic used in both blocks
Device: Siemens Acuson x300 3-5MHz Ultrasound — Ultrasound used to aid in the blocks

SUMMARY:
The purpose of this study to compare erector spinae block to transversus abdominis plane block in bariatric surgeries regarding analgesic efficacy and postoperative oxygenation and respiratory complications

DETAILED DESCRIPTION:
The erector spinae plane (ESP) block is an interfascial block proposed to provide analgesia for chronic pain and perioperative period. it can provide both visceral and somatic abdominal analgesia if the injection were performed at a lower thoracic level. ESP block is effective, easy to perform, and can be performed in a short time. Therefore, bilateral ESP block may have comparable or improved analgesic effect in upper and lower abdominal surgical procedures when compared to other suitable plane blocks.

Transversus abdominis plane (TAP) block technique is to reduce postoperative pain and is a part of current analgesic regimen for many abdominal surgeries . Moreover, it was found that posterior TAP block appears to produce more prolonged analgesia than the lateral TAP block. Ultrasound guided TAP block is a feasible, minimally invasive technique . It reduces the postoperative requirement of opioid analgesics, decreases the incidence and severity of postoperative nausea and vomiting, improves patient satisfaction, and allows early readiness for discharge postoperatively.

Both blocks is effective in reducing postoperative complication and need of analgesia , To our knowledge there is no comparative study between the two blocks to this population .

the investigators aim to compare the perioperative analgesic effect between TAP block and ES block in bariatric .

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18 <60
* Obese patients ; Body mass index(BMI) 40-50 kg/m2
* Both sexes
* American Society of Anesthesiologists(ASA) physical status classes II and III
* Patients scheduled for laparoscopic bariatric surgery i.e. sleeve gastrectomy and/or Roux-en-Y gastric bypass (RYGB)surgeries

Exclusion Criteria:

* Refusal of regional block
* Patients with neurological, psychological disorders or those lacking cooperation
* Patients scheduled for concomitant laparoscopic cholecystectomy or paraumbilical hernia repair or those with history of previous bariatric surgery or obstructive sleep apnea
* Patients with anatomic abnormalities at site of injection, skin lesions or wounds at site of proposed needle insertion.
* Patients with bleeding disorders defined as (INR >2) and/ or (platelet count <100,000/µL)
* Patients with hepatic disease e.g. liver cell failure or hepatic malignancy or hepatic enlargement.
* Patients who are allergic to amide local anesthetics.
* Cases converted to open surgery will also be excluded from the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
efficacy of block | first 24 hours postoperative
  The analgesic efficacy of erector spinae block versus TAP block assessed by visual analogue score(range from 1 denoted the least pain to 10 as the worst pain) in 24hr in laparoscopic bariatric surgery.

SECONDARY OUTCOMES:
failure rate | first hour postoperatively
  Failure rate in both groups

OTHER OUTCOMES:
feasibility of block | preoperative
  Time taken to perform a successful block
ambulation | 24 hour
  Time to ambulate in both groups
arterial oxygen tension to fraction of inspired oxygen ratio | 12, 24 hours postoperative
  p/f ratio after first 12 , 24 hours postoperatively in both groups
pulmonary complications | 12,24 hours postoperative
  Incidence of postoperative pulmonary complication ( chest x-ray at 12, 24 hr postoperative )

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tulgar S, Selvi O, Kapakli MS. Erector Spinae Plane Block for Different Laparoscopic Abdominal Surgeries: Case Series. Case Rep Anesthesiol. 2018 Feb 18;2018:3947281. doi: 10.1155/2018/3947281. eCollection 2018. PMID 29670771
- [Background] Abdallah FW, Laffey JG, Halpern SH, Brull R. Duration of analgesic effectiveness after the posterior and lateral transversus abdominis plane block techniques for transverse lower abdominal incisions: a meta-analysis. Br J Anaesth. 2013 Nov;111(5):721-35. doi: 10.1093/bja/aet214. Epub 2013 Jun 27. PMID 23811424
- [Background] Mittal T, Dey A, Siddhartha R, Nali A, Sharma B, Malik V. Efficacy of ultrasound-guided transversus abdominis plane (TAP) block for postoperative analgesia in laparoscopic gastric sleeve resection: a randomized single blinded case control study. Surg Endosc. 2018 Dec;32(12):4985-4989. doi: 10.1007/s00464-018-6261-6. Epub 2018 Jun 4. PMID 29869078